CLINICAL TRIAL: NCT02018380
Title: Immediate Effects of Shock Absorbing Insoles on Knee Pain, Functional Mobility, and Lower Extremity Biomechanical Characteristics in Persons With Knee Osteoarthritis
Brief Title: Effects of Shock Absorbing Insoles on Knee Pain and Walking in Persons With Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Winston Salem State University (Other)
Collaborators: Wake Forest University Health Sciences (Other); University of North Carolina (Other)
Responsible Party: Principal Investigator, Judy L. Foxworth, PT, PhD, OCS, Associate Professor, Winston Salem State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2986-06-0038
Record Dates: First submitted 2009-06-29; First posted 2013-12-23 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Shock Absorbing Insoles vs. Athletic shoes (Experimental)
  Interventions: Other: Shock Absorbing Insole (SofSole Athletes Plus)

INTERVENTIONS:
Other: Shock Absorbing Insole (SofSole Athletes Plus) — The shock absorbing insole used in this study was the SofSole Athletes Plus, (Implus Inc, Durham, NC), recommended by the manufacturer for repetitive activities such as running and walking. It is readily available in most athletic shoe stores, retailing for under $20.00. The insole is full-length with a curved last made of Implus XP that has a shore A durometer reading of 60 (0 = softest to 100 = hardest).
  Other Names: SofSole Athletes Plus

SUMMARY:
Osteoarthritis (OA) is a progressive, chronic disease affecting more than 20 million Americans. There is no known cure for OA and management includes pain control and prevention of functional decline.

Purpose: To investigate the immediate effects of a shock absorbing insole (SAI) placed in the shoe on knee pain, functional mobility and lower extremity biomechanics.

DETAILED DESCRIPTION:
Sixty adults (age 50+) with knee OA and pain will be recruited. A physician will diagnose the severity of knee OA through radiographs. Participants will be tested in the KBR Human Performance Lab on the campus of Winston Salem State University (WSSU). Participants will complete a demographic form and a survey about their knee pain and function. Participants will be evaluated under two conditions: 1) with SAI placed inside the shoe and 2) shoes alone. There are three walking tasks: 1) walking 25 feet at their usual pace; 2) walking 25 feet at a fast pace; 3) walking six minutes for distance; and a 4) biomechanical gait analysis. After each of the walks, participants will rate the amount of knee pain they experienced. During the biomechanical analysis, participants will walk down a 20 foot walkway while wearing reflective markers. Eight cameras and a force plate embedded in the walkway will measure the amount of body movement and the forces applied to the leg joints during walking.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older
* Radiographic evidence of knee OA in the test extremity (K-L grading scale = 1 to 4)
* Knee pain (WOMAC pain subscore of 4 or more and report moderate pain on at least 1 listed activity in the WOMAC) on most days
* Able to speak, write, and understand English
* Able to walk 25 feet without an assistive device
* Must wear a shoe size available in the lab (Women's 6-10 and Men's 8-14)
* Able to attend two sessions of data collection within 14 days

Exclusion Criteria:

* Currently wearing some type of foot orthosis (custom or over-the counter)
* Had lower extremity surgery of the test leg in the past 12 months
* Had a total knee replacement on the involved leg
* Had hip and/or ankle OA in the involved leg
* Had a neuromuscular disease disorder which affected their walking ability

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-08; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Knee pain while walking | Baseline

SECONDARY OUTCOMES:
Ground Reaction Forces | Baseline
Knee joint kinetics during stance phase of gait | Baseline
Gait speed | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Judy L Foxworth, PT, PhD, Principal Investigator — Winston Salem State University; Darin Padua, ATC, PhD, Study Chair — Unversity of North Carolina; Stephen Messier, PhD, Study Director — Wake Forest University
Locations (1):
- Winston Salem State University, Winston-Salem, North Carolina, United States